CLINICAL TRIAL: NCT04262986
Title: A Brief Motivational Enhancement Lifestyle Modification Programme to Reduce Body Weight in Overweight Subjects With OSA: Needs Assessment
Brief Title: A Brief Lifestyle Modification Programme in Overweight Subjects With Obstructive Sleep Apnoea - Needs Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant Professor, The University of Hong Kong
Other Study IDs: UW 20-068-1
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnoea; Overweight
Keywords: Lifestyle modification; Obstructive sleep apnoea; Overweight
MeSH Terms: conditions — Sleep Apnea, Obstructive; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea (OSA) is a common chronic disease and associated with cardiovascular and neurocognitive sequelae. Overweight is a common, reversible risk factor of OSA, and the rapid rise in obesity worldwide may lead to increases in OSA and related adverse health outcomes. Weight-loss interventions, especially comprehensive lifestyle interventions, are associated with improvements in OSA severity, cardiometabolic comorbidities, and quality of life. However, the intensive nature of these programmes often pose a barrier to adherence. Furthermore, although there is strong evidence to support the value of mobile text messaging to promote physical activity and healthy eating in clinical and community settings, messaging has rarely been applied in interventions for overweight OSA subjects.

The proposed study aims to examine the feasibility of a brief lifestyle modification programme that makes use of smartphone technology (WhatsApp or WeChat) to empower subjects to start doing simple and easy-to-do exercises that can be easily integrated into daily life for gradual lifestyle change.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common chronic disease and associated with cardiovascular and neurocognitive sequelae. Overweight is a common, reversible risk factor of OSA, and the rapid rise in obesity worldwide may lead to increases in OSA and related adverse health outcomes. Weight-loss interventions, especially comprehensive lifestyle interventions, are associated with improvements in OSA severity, cardiometabolic comorbidities, and quality of life. However, non-adherence is commonly seen in such lifestyle modification programmes. Such programmes are often intensive and pose a barrier to adherence. Researchers have suggested that programmes with fewer sessions may improve the completion rates. As yet, there have been no randomised trial assessing the feasibility and effectiveness of a brief theory-based lifestyle modification programme.

Furthermore, although there is strong evidence to support the value of mobile text messaging to promote physical activity and healthy eating in clinical and community settings, messaging has rarely been applied in interventions for overweight OSA subjects. In Hong Kong, where smartphone penetration is extensive (89% in 2017), utilising messaging as an intervention tool may be especially valuable.

The proposed study will examine the perceived burden and informational needs and preferences of overweight subjects with OSA, especially in relation to physical activity. The study will also examine the feasibility of a brief lifestyle modification programme that makes use of smartphone technology (WhatsApp or WeChat) to provide personalised support and empower subjects to start doing simple and easy-to-do exercises that can be easily integrated into daily life for gradual lifestyle change and weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above;
* Performed sleep test in sleep laboratory; and
* Mentally fit to provide informed consent and answer self-administered questionnaire.

Exclusion Criteria:

* Those on CPAP or oral appliance treatment;
* Diagnosed with psychiatric illness; or
* Unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with obstructive sleep apnoea
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Preference on physical activity | Immediately after obtaining written consent
  Outcome-based questions with categorical choices

SECONDARY OUTCOMES:
Current physical activity practices | Immediately after obtaining written consent
  Outcome-based questions with categorical choices
Preference on programme contents and information | Immediately after obtaining written consent
  Outcome-based questions with categorical choices
Preference on m-Health information | Immediately after obtaining written consent
  Outcome-based questions with categorical choices
Daytime Sleepiness | Immediately after obtaining written consent
  Epworth Sleepiness Scale, ranged from 0 - 24 scores. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life. Score >10 is interpreted as excessive daytime sleepiness
Sleep quality | Immediately after obtaining written consent
  A single-item sleep quality scale; range from 0 -10; Higher score is interpreted as better sleep quality
Dietary consumption habits | Immediately after obtaining written consent
  Outcome-based questions with categorical choices

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Subject consent did not include sharing personal information to other researchers.

REFERENCES:
- [Background] Dobrosielski DA, Papandreou C, Patil SP, Salas-Salvado J. Diet and exercise in the management of obstructive sleep apnoea and cardiovascular disease risk. Eur Respir Rev. 2017 Jun 28;26(144):160110. doi: 10.1183/16000617.0110-2016. Print 2017 Jun 30. PMID 28659501
- [Background] Hudgel DW, Patel SR, Ahasic AM, Bartlett SJ, Bessesen DH, Coaker MA, Fiander PM, Grunstein RR, Gurubhagavatula I, Kapur VK, Lettieri CJ, Naughton MT, Owens RL, Pepin JL, Tuomilehto H, Wilson KC; American Thoracic Society Assembly on Sleep and Respiratory Neurobiology. The Role of Weight Management in the Treatment of Adult Obstructive Sleep Apnea. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 15;198(6):e70-e87. doi: 10.1164/rccm.201807-1326ST. PMID 30215551
- [Background] Hall AK, Cole-Lewis H, Bernhardt JM. Mobile text messaging for health: a systematic review of reviews. Annu Rev Public Health. 2015 Mar 18;36:393-415. doi: 10.1146/annurev-publhealth-031914-122855. PMID 25785892
- See also: HKSAR Thematic Household Survey: Personal computer and Internet penetration — https://www.statistics.gov.hk/pub/B11302642018XXXXB0100.pdf